CLINICAL TRIAL: NCT03541083
Title: Blinatumomab Added to Prephase and Consolidation Therapy in Precursor B-acute Lymphoblastic Leukemia in Adults. A Phase II Trial
Brief Title: Blinatumomab Added to Prephase and Consolidation Therapy in Precursor B-acute Lymphoblastic Leukemia in Adults.
Acronym: HOVON146ALL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO146; 2017-000766-30 (EudraCT Number)
Record Dates: First submitted 2018-03-20; First posted 2018-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: ALL, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab (Experimental): After a 5-day steroid prephase patients will receive two weeks continuous infusion of blinatumomab. Then the first remission-induction course will be given after one week interruption. Subsequent therapy with 4 cycles of chemotherapy and two 4-week courses of blinatumomab will follow, and subsequently depending on risk group, eligibility and a suitable donor either allogeneic stem cell transplantation or 2 year maintenance treatment.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — prephase and consolidation (I and II)
  Other Names: Blincyto

SUMMARY:
Blinatumomab is a new active bispecific monoclonal antibody for treatment of lymphoid malignancies, including ALL (acute Lymphoblastic Leukemia ) whose activity for remission induction needs to be explored in combination with standardized treatment in order to improve outcome of this disease which is still lethal in most adult patients. Ultimate proof of efficacy resides in an increase of reaching MRD ( minimal residual disease) negativity, prolongation of that response, and long-term survival. Since hematological response rate in adult ALL is high already and defining long-term survival in a large clinical trial takes many years, this trial aims to improve the strength of the MRD response as defined by achieving complete MRD negative response (ie, < 10^-4) after the first consolidation phase including blinatumomab. This MRD response will be assessed by Real-Time Quantitative Polymerase Chain Reaction (RQ-PCR) analysis of patient-specific Ig/TCR (T-cell receptor ) gene rearrangements. When MRD data are missing, MRD positivity will be assumed. Although younger (up to 40 years of age) patients are treated more intensively than older patients (older than 40 years of age), the investigational questions concerning blinatumomab can be examined in both subgroups as both younger and older patients receive the same type of chemotherapy courses with dose adjustments for chemotherapeutic agents only for patients above 60 years of age.

DETAILED DESCRIPTION:
This trial aims to improve the strength of the MRD ( minimal residual disease) response as defined by achieving complete MRD negative response (ie, < 10^-4) after the first consolidation phase including blinatumomab.

ELIGIBILITY:
Inclusion Criteria:

* Primary CD19 (cluster of differentiation antigen 19) positive precursor B-ALL (excluding mature B-cell ALL and B-lymphoblastic lymphoma, but including Philadelphia positive/BCR-ABL (Abelson murine leukemia viral oncogene homolog 1) positive ALL) and CD19 positive mixed phenotype acute lymphoblastic leukemia (MPAL);
* Patients aged 18 to 70 years inclusive;
* WHO ( World Health Organization) performance status 0-2;
* Negative pregnancy test at inclusion, if applicable;
* Written informed consent;
* Patient is capable of giving informed consent.

Exclusion Criteria:

* Mature B-cell leukemia/lymphoma, B-lymphoblastic lymphoma, isolated extramedullary disease;
* CML (Chronic myeloid leukemia) in blast crisis;
* Acute undifferentiated leukemia;
* Previous treatment with chemotherapy for precursor B-ALL (maximum 5 days of steroid treatment is allowed)
* Persistent liver enzyme disorders (ASAT/ALAT) >5xULN (Upper Limit of Normal) despite steroid pre-treatment (see also 8.1.3.)
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease);
* Severe pulmonary dysfunction (CTCAE grade III-IV, see appendix D);
* Severe neurological or psychiatric disease;
* Active, uncontrolled infection;
* Clinically overt central nervous system disease;
* History of active malignancy during the past 5 years with the exception of basal cell carcinoma of the skin or stage 0 cervical carcinoma;
* Patient known to be HIV-positive;
* Pregnant or breast-feeding female patients;
* Unwilling or not capable to use effective means of birth control (all men, all premenopausal women under the age of 50 need contraception for two years after the last period, and women older than 50 years for at least one year);
* Current participation in another clinical trial;
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients that achieve MRD ( minimal residual disease) negative response, measured by Polymerase Chain Reaction (PCR), after the first blinatumomab consolidation course. MRD negative response is defined as MRD <10-4 | 1 year after closure of study

SECONDARY OUTCOMES:
Complete and molecular response rate following induction and after blinatumomab consolidation ll by the addition of i.v. blinatumomab to standard prophase, consolidation and intensification therapy | 1 year after closure of study
Event-free survival (EFS) | 1 year after closure of study
Relapse-free survival (RFS) | 1 year after closure of study
Overall survival (OS) | 1 year after closure of study
Adverse events; assessing the safety and toxicity of adding blinatumomab to standard prophase and consolidation therapy (two times) in adult ALL | 1 year after closure of study
RFS and OS from start allogeneic transplantation and from start maintenance RFS | 1 year after closure of study
Comparison of molecular and flowcytometric MRD measurements at the same timepoints | 1 year after closure of study

CONTACTS AND LOCATIONS:
Overall Officials: A.W. Rijneveld, Dr., Principal Investigator — Erasmus MC, Rotterdam
Locations (18):
- Belgium (6):
  - BE-Antwerpen Edegem-UZA, Antwerp
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Brugge-AZBRUGGE, Bruges
  - BE-Gent-UZGENT, Ghent
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Roeselare-AZDELTA, Roeselare
- Netherlands (12):
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The foundation of Hemato-Oncologie voor Volwassenen Nederland (HOVON - the Haemato Oncology Foundation for Adults in the Netherlands). — http://www.hovon.nl